CLINICAL TRIAL: NCT06448910
Title: Lung-AK104 Study: Cadonilimab(AK104) Plus Concurrent Chemoradiotherapy in Patients With Locally Advanced, Unresectable, Stage Lll Non-Small Cell Lung Cancer
Brief Title: Cadonilimab(AK104) Plus Concurrent Chemoradiotherapy in Patients With Locally Advanced, Unresectable, Stage III NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lung-AK104
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: NSCLC; Locally Advanced Lung Carcinoma
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadonilimab plus concurrent chemoradiotherapy (Experimental)
  Interventions: Drug: Cadonilimab (AK104)

INTERVENTIONS:
Drug: Cadonilimab (AK104) — Participants will receive 2 cycles of induction therapy with cadonilimab combined with carboplatin/cisplatin plus etoposide, followed by standard concurrent chemoradiotherapy (thoracic radiotherapy + carboplatin/cisplatin plus etoposide), and finally consolidation therapy with cadonilimab (AK104) for 1 year.
  Other Names: Concurrent Chemoradiotherapy

SUMMARY:
The goal of this single arm, phase II clinical trial is to evaluate the efficacy and safety of cadonilimab (AK104) as induction and consolidation therapy in locally advanced/unresectable non-small cell lung cancer (NSCLC) patients treated with concurrent chemoradiotherapy.

Participants will receive 2 cycles of induction therapy with cadonilimab combined with carboplatin/cisplatin plus etoposide, followed by standard concurrent chemoradiotherapy (thoracic radiotherapy + carboplatin/cisplatin plus etoposide regimen chemotherapy), and finally consolidation therapy with cadonilimab (AK104) for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old;
* ECOG physical status: 0-1;
* The expected survival time is more than 3 months;
* Patients with locally advanced/unresectable stage IIIA-C NSCLC confirmed by histopathology or cytology based on the AJCC 8th edition staging system at initial diagnosis；
* Did not receive any anti-tumor treatment;
* No known sensitive EGFR/ALK/ROS1 mutations
* According to RECIST criteria, at least one measurable lesion must be used as the target lesion
* Good organ function ≤ 7 days before the first dose of study drug, as indicated by the following laboratory values:

  1. Absolute neutrophil count (ANC) ≥1.5 x 109/L, platelet ≥100 x 109/L, hemoglobin ≥90g/L;
  2. INR or PT ≤1.5 x ULN;
  3. aPTT ≤1.5 x ULN;
  4. Total serum bilirubin ≤1.5 x ULN;
  5. AST and ALT ≤ 2.5x ULN or ≤5×ULN in patients with liver metastases;
  6. albumin ≥25 g/L (2.5 g/dL);
  7. Serum creatinine ≤1.5 times the upper limit of normal value (ULN), or serum creatinine clearance calculated by Cockcroft-Gault formula >50 mL/min;
* Informed consent signed by patients or their legal representatives was obtained, and the study protocol and follow-up procedure were followed.
* Patients of childbearing potential had to be willing to continue using high-potency contraception for the duration of the study and for ≥120 days after the last dose of Cadonilimab (AK104).

Exclusion Criteria:

* Pathological types of mixed small cell and non-small cell lung cancer;
* Patients with known EGFR/ALK/ROS1 mutations;
* Patients have received an approved systemic anticancer therapy or systemic immunomodulatory agent (including, but not limited to, interferon, interleukin-2, and tumor necrosis factor) within 4 weeks before the first dose;
* Have received a live or attenuated live vaccine within 4 weeks before enrollment or are expected to require a live or attenuated live vaccine during the study or within 5 months after the last dose of Cadonilimab (AK104);
* Patients allergic to Cadonilimab(AK104) or any of the ingredients, or the container;
* Untreated patients with chronic hepatitis B or chronic hepatitis B virus carriers with HBV DNA≥500 IU/mL or patients with active hepatitis C:
* Patients with inactive HBsAg carriers and medically stable active HBV infection (HBV DNA<500 IU/mL) were eligible. Only to hepatitis b core antibody (anti HBc antibody) patients who tested positive for HBV DNA testing.
* Patients who were negative for hepatitis C virus (HCV) antibodies at screening or who were positive for HCV antibodies at screening and subsequently tested negative for HCV RNA were eligible. HCV RNA testing will be performed only in patients who are positive for hepatitis C virus (HCV) antibodies.

Note: the hepatitis b surface antigen (HBsAg) can be detected or patients with HBV DNA can be detected, should according to the guidelines for treatment. Patients receiving antiviral treatment at screening were supposed to have been on treatment for more than 2 weeks before enrollment and to have continued treatment for 6 months after discontinuation of the study drug.

* Need systemic treatment of active autoimmune disease, the researchers reckon have an impact on research and treatment of patients;
* Any condition requiring systemic treatment with a corticosteroid (prednisone or equivalent >10 mg/ day) or other immunosuppressive agent, within 14 days before the first dose of the study drug, that was assessed by the investigator as having an impact on the study treatment;
* Severe chronic or active infection (including tuberculosis infection, etc.) requiring antimicrobial, antifungal, or antiviral systemic therapy within 14 days prior to the first dose of study drug
* Always allogeneic stem cell transplantation or organ transplantation;
* Meet the following any kind of cardiovascular risk factors of standard:

  1. Cardiogenic chest pain ≤28 days before the first dose of study drug, defined as moderate pain that limits instrumental exercise of daily living;
  2. Symptomatic pulmonary embolism ≤28 days before the first dose of study drug;
  3. Any history of acute myocardial infarction ≤6 months before the first dose of study drug;
  4. Any history of New York Heart Association (NYHA) class III or IV heart failure ≤6 months before the first dose of study drug;
  5. Any ventricular arrhythmic event of grade ≥2 occurred ≤6 months before the first dose of study drug.
  6. History of any cerebrovascular accident ≤6 months before the first dose of study drug;
  7. Corrected QT interval (QTc) (corrected with Fridericia's method) >450 msec; Note: If the QTc interval on the initial ECG was >450 ms, a subsequent ECG was performed to rule out the result
  8. Left ventricular ejection fraction (LVEF) ≤ the lower limit of normal (LLN) as assessed by echocardiography (ECHO);
  9. Any syncope or seizure occurring ≤28 days before the first dose of study drug;
* Patients with uncontrolled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg);
* Bleeding, thrombotic disorders, or use of an anticoagulant (e.g., warfarin) or similar medication requiring therapeutic INR monitoring within 6 months before the first dose of a study drug that, in the investigator's judgment, may have influenced treatment;
* Patients with any sign or history of bleeding that was assessed by the investigator as having an impact on the study protocol; Patients who had any bleeding event of grade 3 or higher, nonhealed wound, ulcer, or fracture within 4 weeks before the first dose;
* Hemoptysis > 50ml/d;
* The central cavity or tumor was shown to invade or be adjacent to large vessels by imaging studies, and the tumor was assessed by the investigator as likely to invade large vessels and cause fatal bleeding.
* Unable to swallow capsules or significant influence disease or a history of gastrointestinal function, such as malabsorption syndrome, stomach or intestinal resection, bariatric surgery, with symptoms of inflammatory bowel disease, or incomplete or complete intestinal obstruction.
* Patients requiring treatment with gastric ph-regulating drugs, including proton pump inhibitors and/or H2 antagonist drugs. Patients can convert antacids;
* Patients with a history of uncontrolled systemic diseases, including diabetes mellitus, hypertension, pulmonary fibrosis, or acute lung disease, that were assessed by the investigator as having an impact on the study treatment;
* Patients with a history of major illness or clinical manifestations that may affect the function of organ systems and are considered by the investigator to have an impact on the study treatment;
* Had undergone any major surgery requiring general anesthesia within 28 days or less before the first dose;
* There are underlying medical conditions or alcohol/drug abuse or dependence that contraindicate the use of the experimental drug or preclude the administration of the study drug, or may affect the interpretation of the results, or place the patient at a high risk of treatment complications;
* Known human immunodeficiency virus (HIV) infection;
* Any activity before the group 2 years or less malignant tumor, except in the study of the specific cancer and any local recurrence has been cured of cancer (such as removal of basal cell or squamous cell cancer, superficial bladder cancer, cervical or breast carcinoma in situ);
* Pregnant or lactating women, or male and female patients who plan to have a child during the study period;
* Participate in another therapeutic clinical study at the same time, unless it is an observational (nonintervention) clinical study or is in the follow-up period of an intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate，ORR | 3 years
  According to RECISIT1.1 criteria, the proportion of patients achieving CR and PR as their best response before initial disease progression was evaluated.
The incidence rate of treatment-related adverse events | 3 years
  The proportion of treatment-related toxicity to the total number of evaluable cases was evaluated according to CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
ORR before Concurrent Chemoradiotherapy | 3 years
  Objective response rate was evaluated according to RECIST 1.1 criteria after two courses of Cadonilimab combined with EP chemotherapy and before the start of concurrent chemoradiotherapy
disease control rate before Concurrent Chemoradiotherapy | 3 years
  Disease control rate was evaluated according to RECIST 1.1 criteria after two courses of AK104 combined with EP chemotherapy and before the start of concurrent chemoradiotherapy
Overall survival，OS | 3 years
  The time from enrollment to death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.
Progression free survival，PFS | 3 years
  The time from enrollment to disease progression or death from any cause. Patients who were still alive at the time of analysis will have the date of their last contact as the cutoff date.
12 months PFS | 3 years
  The proportion of patients who had progression or died from any cause from the first day of enrollment through 12 months among all participants who received at least one dose of Cadonilimab.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No